CLINICAL TRIAL: NCT04196751
Title: An Evaluation Study to Identify the Effectiveness of Clinical Supervision With Regards to Work-related Strain, Sense of Coherence, Increased Cultural Sensitivity and the Impact on Patient's Care: A Prospective Longitudinal Study in Mental Health Services in Qatar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MRC-01-18-409
Record Dates: First submitted 2019-07-24; First posted 2019-12-12 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Work Related Stress; Sense of Coherence; Cultural Sensitivity; Clinical Supervision
Keywords: clinical supervision, work related stress, sense of coherence, cultural sensitivity, mental health nursing
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Intervention Model Description: Open-label Prospective Longitudinal Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Supervision Intervention (Experimental): All the enrolled participants will be undergoing Clinical Supervision sessions with their selected supervisors for pre-identified objectives for their skill and knowledge development.
  Interventions: Other: Clinical Supervision

INTERVENTIONS:
Other: Clinical Supervision — After baseline data collection, participants will be invited to attend training on clinical supervision (CS). Education will be delivered in 3 phases. 1-Orientation to the CS model 2-Integration of theory into practice and 3-Skill advancement for supervisors. After training, participants will be encouraged to choose a supervisor, identify objectives for skill development. They will be advised to meet their supervisor once a month for 60 minutes (Due to COVID 19 pandemic the participants can have either one-to-one session in-person or virtually (Microsoft Team), however, if the supervisor and the supervisee working in the same campus can have their one-to-one session as per their preferences. Supervisor-supervisee will be working together to achieve the stated goals. Only the recorded attendance and nature of the session will be used for research purpose. Data will be collected at baseline, 6&12 month with pre-specified tools.

SUMMARY:
Clinical supervision (CS) is a pragmatic approach, which enables nurses to work together; it can create a positive nursing environment, reduce stress, and increase clinical skills through peer support. Previous research has demonstrated its positive effects on nurses wellbeing, sense of coherence, and professional accountability. However, there is lack of evidence for its influence on cultural sensitivity.

The Qatar National Health Strategy (Ministry of Public Health, 2018) and the Qatar National Mental Health Strategy (Supreme Council of Health, Qatar, 2013) have both given significant importance on building the health workforce capacity to meet the growing needs of the population. Aligning with these strategies, Hamad Medical Corporation (HMC) Mental Health Service's Executive Committee has taken a decision to implement clinical supervision to develop a supporting framework to strengthen the professional skills of the nursing workforce. In order to implement it efficiently, guidelines and education curriculum have been developed. The aim of the study is to evaluate the implementation of CS. In addition, investigators will also explore the impact of clinical supervision on the work-related strain, sense of coherence, cultural sensitivity and the impact on patient care. A longitudinal approach will be adopted using pre and post-testing. The required power sample size is calculated to be 136 nurses. Enrolled participants will receive an educational programme regarding clinical supervision and will be requested to choose a supervisor based on their learning requirements. Through the clinical supervision process, supervisee self-reflection, facilitated by the supervisor. The supervisor will, in addition, enable opportunities for professional growth by the sharing of skills and knowledge in relation to particular clinical challenges. In addition, they will also provide opportunities for emotional restoration through the exploration of stressful issues that have occurred in the workplace.

Participants will be scheduled to engage in one to one sessions with their supervisor once a month for an hour. The study will be conducted for 18 months (2 months for baseline data collection, 2 months for educational preparation, 12 months of intervention and lastly 2 months for post-intervention data collection) from the date of the participant's enrollment. The outcome measures include the sense of coherence, work-related strain, cultural sensitivity, the total number of nurse instigated Occurrence, Variance and Accident (OVA) initiated during the course of this study and the efficacy of clinical supervision sessions. Data will be collected before education sessions are delivered (baseline), at 6th month and at the 12th month. The investigators will use the Statistical Package for the Social Sciences (SPSS) and STATA for analysis. The study may identify an effective way of reducing work-related strain and enhancing the sense of coherence, cultural sensitivity, and quality of patient care.

ELIGIBILITY:
Inclusion Criteria:

* Licensed nursing staffs (QCHP) with grade 107 and above will be invited to participate in the study.

Exclusion Criteria:

* Staff who are on extended leave.
* New staff under preceptorship.
* Staff who do not wish to participate in the research project.
* Unlicensed nursing professionals (e.g. nursing aid).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Work-related Strain | At baseline, and then at 6th month and 12th month after the first clinical supervision session
  The literature suggests that work-related stress and injuries are more common among nurses. Clinical supervision aims to provide support to nurses and guide them to identify their learning needs, improve their knowledge and skills to deal with complex situations and subsequently may reduce work-related strain. To assess the effectiveness of clinical supervision on the work-related strain, investigators will use the Work-Related Strain Inventory (WRSI). It consists of 18 statements designed to measure the feelings of psychological strain in occupational settings. The possible scores for the WRSI range from 18-72, the higher the score, the stronger the feelings of experiencing work-related strain. Data on WRSI will be collected at baseline (before Clinical Supervision sessions), at 6th and 12th month after the first clinical supervision session. The change in the mean scores will be assessed using an appropriate statistical test.
Sense of Coherence | At baseline, and then at 6th month and 12th month after the first clinical supervision session
  A high sense of coherence is a pre-requisite for successful adaptation to a stressful situation- which leads to better health and wellbeing. Investigators will use a short form with 13 items of Sense of Coherence. These 13 items comprise three components: comprehensibility, manageability, and meaningfulness. The respondents indicate agreement or disagreement on a seven category semantic differential scale with two anchoring responses tailored to the content of each item. Five items (1,2,3,5, and 7) needs to be reversed before summing the total scores. The total score can range from 13 to 91, and a higher score indicates higher Sense Of Coherence. Data on SOC will be collected at baseline (before intervention), at 6th and 12th month after the first clinical supervision session. The change in the mean scores will be assessed using an appropriate statistical test.
Intercultural Sensitivity | At baseline, and then at 6th month and 12th month after the first clinical supervision session
  The majority of the nursing workforce in Qatar is of expatriates. Studies show that migrant nurses often face language barriers, cultural diversity, and lack of trust and mutual respect. In this study, investigators are anticipating that supervisee and supervisor may be from different cultures. It is expected that this may promote mutual respect and cultural sensitivity. Intercultural Sensitivity Scale (ICS) will be used to assess cultural sensitivity. The ICS is subdivided into five subscales, and these are Interaction Engagement, Respect for Cultural Differences, Interaction Confidence, Interaction Enjoyment and Interaction attentiveness. A high score indicated higher Intercultural Sensitivity. Data on ICS will be collected at baseline, at 6th and 12th months after the first session of clinical supervision. The change in the mean scores will be assessed.
Perceived effectiveness of Clinical Supervision | After the 12th month from the first session of clinical supervision session.
  Clinical supervision is widely accepted as being a good thing, but until now, this has been more a statement of faith rather than fact. Manchester Clinical Supervision Scale-26 (MCSS-26) will be used to understand the key elements of clinical supervision from the supervisees' perspective. The Manchester Clinical Supervision Scale is designed to establish its true merits once and for all. Investigators using the MCSS with 26 items with six subscales on the five-point Likert scale ranging from '0-strongly disagree' to '4-strongly agree' with a higher score indicating effectiveness. This version is widely tested in a number of studies. The six subscales are: importance/value of clinical supervision, finding the time, trust/rapport, supervisor advise/support, improved care/skills, reflection. Data using MCSS-26 will be collected at the end of the 12th month after the first Clinical Supervision session record date.

SECONDARY OUTCOMES:
Correlation between baseline work-related strain, intercultural sensitivity and sense of coherence. | 6 months from the date of enrollment in the study.
  The investigators are aiming to find the correlation between baseline work-related strain, cultural sensitivity and sense of coherence. Total scores of scales and subscales will be explored for the correlation. If the data follows normal deviation, Pearson correlation coefficient will be used. If data follows the non-normal deviation, then the Spearman Correlation coefficient will be used. The test will be used to find the correlation between baseline work-related strain, cultural sensitivity and sense of coherence.
Effect of clinical supervision on the quality of patient care. | 12 months from the initiation of first session of clinical supervision.
  Through this study, investigators will explore the effect of clinical supervision on the quality of care. (The total number of Occurrence Variance and accidents (OVAs) initiated during the study period (December 2019 to December 2020) will be compared with the retrospective cohort of OVAs initiated from December 2017- December 2018).
Association between clinical supervision experience (using MCSS-26) and participants demographic variables. | 12 months from the initiation of first session of clinical supervision.
  To find the association between perceived clinical supervision experience (MCSS-26) and participants demographic variables including age, gender, and other related variables such as highest academic qualification, total years of clinical experience, number of countries worked as a health care professional, current practising unit, nationality, previous exposure to the clinical supervision, method of allocation of supervisor, nationality and grade of supervisor, setting of clinical supervision, and current job grade of supervisee and supervisor, supervisor and supervisee from the same unit. There is no unit for the tool; investigators will sum-up the total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Mental Health Services, Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonge H, Buus N. Exploring Organizational Barriers to Strengthening Clinical Supervision of Psychiatric Nursing Staff: A Longitudinal Controlled Intervention Study. Issues Ment Health Nurs. 2016 May;37(5):332-43. doi: 10.3109/01612840.2016.1154119. Epub 2016 Apr 14. PMID 27077399
- [Background] Antonovsky, A., 1987. Unravelling the mystery of health: How people manage stress and stay well. Jossey-Bass, San Francisco
- [Background] Saxby C, Wilson J, Newcombe P. Can clinical supervision sustain our workforce in the current healthcare landscape? Findings from a Queensland study of allied health professionals. Aust Health Rev. 2015 Sep;39(4):476-482. doi: 10.1071/AH14183. PMID 25725704
- [Background] Chen, G.-M., Starosta, W.J., 2000. The Development and Validation of the Intercultural Sensitivity Scale
- [Derived] Badanapurkar A, Nelson D, Nazarene A, Smith KW, Phiri L, Varghese S, Ramapurath S. Work-Related Strain, Sense of Coherence and Intercultural Sensitivity Among Mental Health Nurses in Qatar: A Cross-Sectional Study. Int J Ment Health Nurs. 2025 Feb;34(1):e13403. doi: 10.1111/inm.13403. Epub 2024 Sep 16. PMID 39283020